CLINICAL TRIAL: NCT05955274
Title: Personalizing Behavioral Parent Training: Improving Reach and Outcomes for Families of Children With ADHD
Brief Title: Mobile Behavioral Parent Training for Childhood ADHD: Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34MH128513 (NIH)
Record Dates: First submitted 2023-07-12; First posted 2023-07-21 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mBPT only (Active Comparator)
  Interventions: Behavioral: Mobile Behavioral Parent Training (mBPT)
- mBPT and just-in-time adaptive intervention (Experimental)
  Interventions: Behavioral: Mobile Behavioral Parent Training (mBPT); Behavioral: Just-in-time intervention: Parenting Strategies

INTERVENTIONS:
Behavioral: Mobile Behavioral Parent Training (mBPT) — The mobile phone application includes behavioral parent training content (for example, praise, effective commands, reward systems) delivered in videos, examples, and quizzes that parents/caregivers access.
Behavioral: Just-in-time intervention: Parenting Strategies — Parents will receive prompts via phone that provide parenting suggestions and parenting feedback when they are interacting with their child.
  Arms: mBPT and just-in-time adaptive intervention

SUMMARY:
The goal of the study is to develop and pilot a personalized behavioral parent training intervention for caregivers of children with attention deficit hyperactivity disorder. The behavioral intervention will teach positive parenting through videos and quizzes that caregivers can access through a smartphone application. The program also gives parents and caregivers in-the-moment feedback their use of parenting strategies.

The main questions to answer are:

Is parenting feedback provided by a smartphone application acceptable to caregivers? Is the phone application usable and acceptable to parents and caregivers of children with attention deficit hyperactivity disorder?

In the pilot trial, participants (parents/caregivers) will be randomly assigned to either (1) use the positive parenting intervention phone application (mobile Behavioral Parent Training: mBPT) or (2) use mBPT and receive brief, personalized phone prompts throughout their participation that target parenting behavior and intervention engagement.

ELIGIBILITY:
Inclusion Criteria:

* currently meets Diagnostic Statistical Manual 5 diagnostic criteria for ADHD
* ages 7 -12
* has at least one parent or primary caregiver who is willing to participate and is able to access the intervention at home via smartphone.

Exclusion Criteria:

* N/A

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Intervention Engagement | Through study completion, average of 10 weeks
  Number of mobile BPT sessions completed divided by the total number of sessions available.
Receipt of Prompts | Through study completion, average of 10 weeks
  Percent of prompts sent that were opened within 20 minutes of being sent

SECONDARY OUTCOMES:
Passive Audio Data- Positive Parenting | During the last 1 week of study completion
  Parenting Behavior- Dyadic Parent Child Interaction Coding System, number of labeled praises and unlabeled praises per hour during last week of study.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Children and Families of Western New York, Buffalo, New York, United States